CLINICAL TRIAL: NCT04079985
Title: Animal-assisted Intervention in Geriatric Patients With Chronic Joint Pain and Polypharmacy
Brief Title: AAI in Elderly Patient With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IDIAPJordiGol
Record Dates: First submitted 2019-07-05; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
Keywords: Animal-assisted therapy; Chronic Pain; Elderly; Primary Health Care
MeSH Terms: conditions — Chronic Pain | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Single-centre, two-arm randomized, controlled, open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental Group underwent a therapeutic intervention based on sessions of kinesitherapy , which is defined as a set of "therapeutic procedures that use movement for the treatment and prevention of diseases of the locomotive apparatus". The experimental group also underwent AAT. We conducted a total of 12 weekly sessions of 60 minutes each with 10 participants.
  Interventions: Other: Animal-assisted therapy
- Control Group (Active Comparator): The Control Group underwent a therapeutic intervention based on sessions of kinesitherapy , which is defined as a set of "therapeutic procedures that use movement for the treatment and prevention of diseases of the locomotive apparatus" without the presence of the therapy dog.
  Interventions: Other: Animal-assisted therapy

INTERVENTIONS:
Other: Animal-assisted therapy — The sessions were held in the primary care centre, and had specific objectives agreed in advance by the research team. The sessions had the following schedule: Session 1, lower extremities in sitting position; Session 2, upper extremities in sitting position; Session 3, cervical spine in sitting position; Session 4, dorsal spine in sitting position; Session 5, lumbar spine in sitting position; Session 6, Static Standing and Upper Extremities; Session 7, Static Standing; Sessions 8, 9, 10 and 11, Dynamic Standing; and Session 12, Safety Reinforcement.

SUMMARY:
BACKGROUND: Nowadays, there is a progressive aging of population. Chronic osteoarticular pain is associated to a bigger consumption of medication and a deterioration of life quality in elderly people that could be improved by boosting education for health from Primary Health Care. JUSTIFICATION: The need to develop non pharmacological treatments in order to get better results in people's global care. PURPOSE: To evaluate the effectivity of group intervention, based on Animal Assisted Therapy, on elderly people suffering from chronic osteoarticular pain and poli-medication; regarding decrease of chronic pain, use of analgesics and improvement of life quality. MATERIAL AND METHOD: Randomized clinical trial, two arms, controlled and open-label. Twelve group sessions of kinesiotherapy with the intervention of a therapy dog in the experimental group (EG), carried out in the Primary Health Centre.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* diagnosis of chronic benign joint pain
* polypharmacy (>5 drugs or active ingredients, of which 2 or more had been prescribed for pain)

Exclusion Criteria:

* severe cognitive deterioration (GDS> 5)
* allergy to or fear of animals

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index at 13 weeks | This questionnaire was administered at baseline and at week 13.
  pain (0-20), stiffness (0-8), functional capacity (0-68)

SECONDARY OUTCOMES:
Change from baseline Lattinen test at 13 weeks | This questionnaire was administered at baseline and at week 13.
  Assesses pain and any incapacity caused by pain, as well as its frequency and intensity, the amount of painkillers taken, and whether sleep is disturbed
Change from baseline EuroQoL Health Questionnaire at 13 weeks | This questionnaire was administered at baseline and at week 13.
  Is a generic self-administered instrument for measuring quality of life related to health
Change from baseline Health Assessment Questionnaire at 13 weeks | This questionnaire was administered at baseline and at week 13.
  Is a self-administered questionnaire that assesses one's ability to perform day-to-day activities, as well as functional capacity
Change from baseline Visual Analog Scale at session 1 | This questionnaire was administered at the baseline of session 1 and through session 1 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 2 | This questionnaire was administered at the baseline of session 2 and through session 2 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 3 | This questionnaire was administered at the baseline of session 3 and through session 3 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 4 | This questionnaire was administered at the baseline of session 4 and through session 4 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 5 | This questionnaire was administered at the baseline of session 5 and through session 5 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 6 | This questionnaire was administered at the baseline of session 6 and through session 6 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 7 | This questionnaire was administered at the baseline of session 7 and through session 7 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 8 | This questionnaire was administered at the baseline of session 8 and through session 8 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 9 | This questionnaire was administered at the baseline of session 9 and through session 9 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 10 | This questionnaire was administered at the baseline of session 10 and through session 10 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 11 | This questionnaire was administered at the baseline of session 11 and through session 11 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Change from baseline Visual Analog Scale at session 12 | This questionnaire was administered at the baseline of session 12 and through session 12 completion, an average of 1 hour
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ortega Bravo, PhD, Study Director — IDIAPJgol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Doctoral thesis — https://www.tesisenred.net/handle/10803/385217